CLINICAL TRIAL: NCT06903403
Title: Comparing Front-of-package Nutrient Labels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Jennifer Falbe, Associate Professor, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2295549
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Nutrition Knowledge; Perceptions; Dietary Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- No-label Control (No Intervention): Participants will see packaged food and beverage items with no front-of-package labels (other than any posted by the manufacturer).
- Nutrition Info Percent Daily Value (Experimental): Participants will see packaged food and beverage items displaying front-of-package labels that list "high", "medium", or "low" for saturated fat, sodium, and added sugars. "High" is defined as 20% or more of the Daily Value per serving, "medium" as 6-19%, and "low" as 5% or less. The label will also list the percent Daily Value for each nutrient per serving. The label will have a white background and black text.
  Interventions: Other: Front-of-package label
- Nutrition Info with Red "High" (Experimental): Participants will see packaged food and beverage items displaying front-of-package labels that list "high", "medium", or "low" for saturated fat, sodium, and added sugars. "High" is defined as 20% or more of the Daily Value per serving, "medium" as 6-19%, and "low" as 5% or less. The label will have a white background and black text, except for the word "high," which will be in white font and highlighted red.
  Interventions: Other: Front-of-package label
- Plain High In (Experimental): Participants will see packaged food and beverage items displaying front-of-package labels that say, "High In [nutrient]" (nutrients: saturated fat, sodium, and/or added sugars) if the item contains 20% or more of the Daily Value per serving for each nutrient. The label will have a white background and black text. If the item is not high in 1 or 2 of the nutrients, the nutrient(s) will not be on the label. If the item is not high in any of the 3 nutrients, the product will not display this label.
  Interventions: Other: Front-of-package label
- Multiple Black Box High In (Experimental): Participants will see packaged food and beverage items displaying front-of-package labels that say, "High In [nutrient]" (nutrients: saturated fat, sodium, and/or added sugars) if the item contains 20% or more of the Daily Value per serving for each nutrient. Each nutrient will have it's own label, a black box with white text. If the item is not high in a nutrient, it will not display the black box label for that nutrient. If the item is not high in any of the 3 nutrients, the product will not display any labels.
  Interventions: Other: Front-of-package label

INTERVENTIONS:
Other: Front-of-package label — Participants will see packaged food and beverage items displayed with labels as specified by their assigned group
  Arms: Multiple Black Box High In; Nutrition Info Percent Daily Value; Nutrition Info with Red "High"; Plain High In

SUMMARY:
The goal of this study is to compare front-of-package labels to a no-label control and to one another: 1.) FDA's Nutrition Info with %DV, 2.) Nutrition Info with red "high", 3.) FDA's High In, 4.) multiple High In labels-one for each nutrient and 5.) a no-label control. Primary outcomes include 1.) correct identification of foods and beverages with the healthiest and least healthy overall nutrient profiles, 2.) perceived healthfulness of products low in two nutrients of concern, and 3.) correct identification of foods and beverages as high in saturated fat, sodium, and added sugars.

DETAILED DESCRIPTION:
The overall goal of this online randomized controlled trial is to compare the performance of FDA's Nutrition Info %DV front-of-package label (FOPL) to a no-label control and other FOPL designs, including the Nutrition Info label without the %DV and with red color for "high in" nutrients, the FDA's High In label, and multiple black box High In labels-one for each nutrient.

The primary outcomes are: 1.) correct identification of foods and beverages with the healthiest and least healthy overall nutrient profiles, 2.) perceived healthfulness of products low in two nutrients of concern, and 3.) correct identification of foods and beverages as high in saturated fat, sodium, and added sugars. Secondary outcomes include: 1.) noticing the nutrition label, 2.) recalling the label's content, 3.) reported use of label when selecting food items, 4.) perceived healthfulness of i.) products not high in any nutrients of concern and ii.) products with different nutrient levels for each nutrient of concern, 5.) selection of a food item high in at least one nutrient of concern for themselves, 6.) selection of a food item high in at least one nutrient of concern for their youngest child (at least 2 years old), 7.) perceived message effectiveness of label for discouraging consumption of foods high in saturated fat, sodium, and added sugars, 8.) time spent on identifying healthiest and least healthy overall nutrient profiles, and 9.) time spent on identifying foods and beverages as high in saturated fat, sodium, and added sugars.

Repeated dichotomous outcomes (e.g., correct selection of healthiest profile, correct selection of least healthy profile, correct identification of product high in nutrients of concern) will be analyzed in mixed effects Poisson regression with robust standard errors. Single dichotomous outcomes (e.g., noticing, use of label, selection of at least one item high in one nutrient of concern) will be analyzed in Poisson regression with robust standard errors. Results will report proportions in each condition and absolute (i.e., percentage point) and relative differences (i.e., probability ratios). Continuous outcomes (e.g., perceived healthfulness, time spent) will be used in linear regression. All regression models will regress the outcome on an indicator for experimental condition. results will report averages by condition and average differential effects between conditions. Analyses will use a two-sided critical alpha of 0.05 to conduct all statistical tests. All confidence intervals presented will be 95% and two-sided. Given the preliminary nature of this study, which is comparing novel FOPLs for the first time, no p-value adjustments for multiple comparisons are planned.

In moderation analyses using interaction terms and stratified models, effect modification of label design on the primary outcomes will be examined by participant nutrition literacy, education, grocery shopping frequency, having children, and type of device used to take the survey.

Additionally, differences in all outcomes between each of the 5 unique conditions will be examined. The modeling approach may be modified if assumptions are not met.

A soft launch of approximately 500 completed surveys will be conducted to verify that the online survey is functioning as intended and to detect any programming errors. There may be another soft launch if any corrections are needed. If the target sample size is not achieved by April 30th, 2025, the data collected thus far will be used in preliminary analysis to provide public comments. The analytic sample will include participants with complete data on the primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Equal or greater than 18 years of age
* English-speaking
* U.S. residents

Exclusion Criteria:

* Failing the attention check question
* Completing the survey in less than one-third of the median completion time (median time calculated when 90% of responses are collected and will be based on the median time of completed questionnaires)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15582 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Correct identification of healthiest profile | Within approximately 5 minutes of intervention exposure
  Participants will view 4 series of 3 products on the same screen, with each product having a nutrient profile. They will be instructed, "Choose the food [beverage] that has the healthiest overall nutrient profile. Consider saturated fat, sodium, and added sugars." Outcome for each series will be dichotomized (1 = correct, 0 = incorrect), and the multiple outcomes will be used in mixed effects Poisson regression with robust standard errors.
Correct identification of least healthy profile | Within approximately 5 minutes of intervention exposure
  Participants will view approximately 4 series of 3 products side-by-side, showing different nutrient profiles. They will be asked "Choose the food [or beverage] with the least healthy overall nutrient profile. Consider saturated fat, sodium, and added sugars." Outcome for each series will be dichotomized (1 = correct, 0 = incorrect) and the multiple outcomes will be used in mixed effects Poisson regression with robust standard errors.
Correct identification of "high" nutrients | Within approximately 5 minutes of intervention exposure
  Participants will view 5 foods and indicate whether each food is high in each of saturated fat, sodium, and added sugars. A "correct" response is identifying a high-in product as high in the corresponding nutrient and identifying a not high-in product as not high in the corresponding nutrient; otherwise the response is "incorrect". The 15 (3 nutrients across 5 products) dichotomous responses will be analyzed in a mixed model, accounting for within subject correlation.
Perceived healthfulness of items low in two nutrients of concern | Within approximately 5 minutes of intervention exposure
  Participants will provide a healthfulness score (response scale from 1-7 ranging from very unhealthy to very healthy) for 4 different products. The score for each product will be used as a continuous outcome in linear regression models.

SECONDARY OUTCOMES:
Noticing the label | Within approximately 5 minutes of intervention exposure
  After a hypothetical shopping task (the first of two shopping tasks), participants will be asked if they noticed any nutrition labels on the food. Analysis will include using the dichotomous outcome of noticing in Poisson regression with robust standard errors.
Recalling the label's content | Within approximately 5 minutes of intervention exposure
  If participants answer "yes" to noticing a nutrition label, they will be asked, "What information was on the label? Select all that apply." Response options will include calories, fiber, saturated fat, sodium, added sugars, cholesterol, protein, calcium, vitamin D, and "none of these". The percent of options correctly selected or not selected will be used in linear regression.
Reported use of label | Within approximately 5 minutes of intervention exposure
  After a hypothetical shopping task (the first of two shopping tasks), if a participant responds "yes" to noticing a label, they will be asked if they used the label when selecting their item. Outcome will be dichotomized and analyzed in Poisson regression.
Perceived healthfulness of (i) items not high in any nutrient of concern and (ii) items with different nutrient levels for each nutrient of concern | Within approximately 5 minutes of intervention exposure
  Participants will provide a healthfulness score (response scale from 1-7) for 5 different products. The score for each product will be used as a continuous outcome in linear regression models.
Selection of a product high in a nutrient of concern for themselves | Within approximately 5 minutes of intervention exposure
  In the second of two shopping tasks, participants will select a food they would purchase for themselves from hypothetical grocery store shelves. The dichotomous outcome is selection of an item that is high in at least one nutrient of concern (compared to not selecting an item high in at least one nutrient of concern), analyzed in Poisson regression with robust SE to directly estimate probability ratios.
Selection of a product high in a nutrient of concern for their child | Within approximately 5 minutes of intervention exposure
  Participants will select a food they would purchase for their youngest child (at least 2 years old) from hypothetical grocery store shelves. The dichotomous outcome is selection of an item that is high in at least one nutrient of concern (compared to not selecting an item high in at least one nutrient of concern), analyzed in Poisson regression with robust SE to directly estimate probability ratios.
Perceived message effectiveness | Within approximately 5 minutes of intervention exposure
  Participants not in the control group will view their assigned label in isolation (i.e., not on a product) and will be asked "How much does this label discourage you from wanting to purchase foods or beverages that are high in saturated fat, sodium, or added sugars?" Response options will range from not at all (1) to a great deal (5). The responses will be treated as a continuous outcome in linear regression.
Time spent on identifying healthiest and least healthy overall nutrient profiles | Within approximately 5 minutes of intervention exposure
  Timer features will be used in the survey to measure the time spent on the primary outcome of identifying healthiest and least healthy overall nutrient profiles. The time (in seconds) will be used as a continuous outcome in linear regression. The top and bottom 2% will be considered outliers and excluded.
Time spent on identifying foods and beverages as high in saturated fat, sodium, and added sugars. | Within approximately 5 minutes of intervention exposure
  Timer features will be used in the survey to measure the time spent on the primary outcome of identifying foods and beverages as high in saturated fat, sodium, and added sugars. The time (in seconds) will be used as a continuous outcome in linear regression. The top and bottom 2% will be considered outliers and excluded.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Falbe, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No